CLINICAL TRIAL: NCT03489096
Title: CryobAllooN Targeting Atrial fibRosIs in Atrial Fibrillation
Acronym: CANARI-AF
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Sponsor-Investigator left the institution
Sponsor: University of Utah (Other)
Collaborators: Medtronic (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB_00109729
Record Dates: First submitted 2018-03-28; First posted 2018-04-05 (Actual); Last update posted 2019-07-19 (Actual); Status verified 2019-07

CONDITIONS: Atrial Fibrillation; Left Atrial Fibrosis
Keywords: Cryoballoon Ablation; Persistent atrial fibrillation; Paroxysmal atrial fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Intervention Model Description: Single-center, open-label pilot study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Cryoballoon Ablation (Experimental): Cryoballoon Ablation: PVI + substrate modification. Left atrial fibrosis ablation in addition to standard pulmonary vein isolation in patients with paroxysmal and persistent atrial fibrillation. Ablation will be performed utilizing the Medtronic Arctic Front Advance Cryoballoon catheter.
  Interventions: Device: Cryoballoon Ablation: PVI + substrate modification

INTERVENTIONS:
Device: Cryoballoon Ablation: PVI + substrate modification — Standard pulmonary vein isolation using cryoballoon ablation, followed by left atrial fibrosis substrate modification using cryoballoon ablation

SUMMARY:
Pulmonary vein isolation (PVI) using cryoballoon ablation is a well-established procedure for the treatment of atrial fibrillation (AF). However, the use of cryoballoon ablation in recent clinical trials have been limited to PVI. As such, patients with paroxysmal AF have been the main recipients of this procedure. In patients with persistent AF, or patients with paroxysmal AF and significant AF substrate other than the pulmonary veins, the utility of cryoballoon ablation is less straightforward. In such patients, the choices are to either use cryoballoon ablation in a PVI-only approach or alternatively, use cryoballoon ablation for PVI followed by the use of radiofrequency ablation for additional ablation and/or substrate modification.

Substrate modification by targeting left atrial fibrosis detected on delayed enhancement magnetic resonance imaging (DE-MRI) is an increasingly popular approach with growing data showing its utility to decrease the risk of recurrence. The ability to use cryoballoon ablation for fibrosis based ablation in addition to PVI will therefore provide a significant advantage.

This study will evaluate feasibility and the outcome of targeted ablation of left atrial fibrosis detected on DE-MRI in addition to pulmonary vein isolation using the Arctic Front Advance Cryoballoon Catheter.

DETAILED DESCRIPTION:
This is a single center open-label pilot study to be performed at the University of Utah Hospital. Patients that are referred for first time ablation of paroxysmal or persistent atrial fibrillation (AF) will be considered to be enrolled in the study. An electrocardiogram (ECG) will be performed at the time of the first clinic visit with the documentation of the rhythm. All patients will be started on an oral anticoagulation (either a novel anticoagulation agent or warfarin with a targeted international normalized ratio (INR) of 2-3). All patients will have a basic metabolic panel, complete blood count, prothrombin time/INR, thyroid-stimulating hormone, and a chest x-ray at the time of the first clinic visit. Women of childbearing potential will have a β-human chorionic gonadotropin test to rule out pregnancy. Within a month prior to the planned ablation, all patients will undergo a DE-MRI to assess pulmonary vein anatomy, fibrosis burden and distribution, and left ventricular function.

All patients will undergo a transesophageal echocardiogram immediately prior to the ablation procedure to rule out thrombus within the left atrial appendage. If thrombus is detected, the procedure will be postponed. AF ablation procedure will consist of pulmonary vein isolation using the Medtronic Arctic Front Advance Cryoballoon Catheter. Following PVI, additional lesions will be placed targeting areas of fibrosis by further manipulation of the catheter from its position within pulmonary vein.

Following ablation, all patients will be observed for 24 hours to assess immediate post procedural complications. All patients will be continued on anticoagulation for at least two months. Patients may be continued on oral anticoagulation beyond two months post-ablation if they are determined to have a high stroke risk profile.

A DE-MRI will be performed on all patients within 24 hours of ablation to assess esophageal thermal injury. Patients with severe esophageal enhancement will have a repeat DE-MRI within 24 hours. Patients with moderate enhancement will have a repeat DE-MRI within 1 week. All patients with persistent esophageal enhancement on repeat DE-MRI will be referred for esophagogastroduodenoscopy. All patients will be placed on a proton pump inhibitor for 1 month.

All patients will be discharged with a 60-day event monitor. Continuation of antiarrhythmic medications will be at the discretion of the performing physician. Following the procedure, a 90-day blanking period will start. Following the blanking period, patients will be monitored for one year for recurrence of AF. Recurrence of AF is defined as a detectable episode of AF, atrial flutter, or atrial tachycardia lasting at least 30 seconds. AF recurrence will be assessed by 30-day event monitors at 3, 6, and 12-months following the blanking period. A chest x-ray will be performed in all patients at the time of their first follow up visit.

All patients will undergo a DE-MRI at 3 months at the time which ablation scar size and burden, progression of left atrial fibrosis as well as presence of pulmonary vein stenosis will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Referred for cryoballoon ablation of paroxysmal or persistent atrial fibrillation
* 18 years of age or older
* Ability to give informed consent in accordance with University of Utah IRB guidelines

Exclusion Criteria:

* Previous ablation for atrial fibrillation or atypical atrial flutter
* Contraindication to MRI contrast agent
* Unquantifiable fibrosis or moderate to severe left-atrial fibrosis (≥ 20%)
* Contraindication for chronic anticoagulation therapy
* Acute coronary syndrome, cardiac surgery, angioplasty, or cerebrovascular disease within the last 2 months
* Implanted cardiac device
* Presence of left atrial thrombus
* Contraindications to cryoballoon ablation including history of cryoglobulinemia, active systemic infection, and presence of one or more pulmonary vein stents
* New York Heart Association (NYHA) class IV heart failure
* Women who are currently pregnant or breast feeding or using unreliable contraceptive measures if premenopausal
* Enrollment in another investigational trial
* Untreated hyperthyroidism or hypothyroidism
* Life expectancy < 12 months due to a terminal disease
* Presence of phrenic nerve injury at baseline elicited by hemidiaphragmatic paralysis on pre-ablation chest x-ray

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-10 (Estimated); Primary Completion 2021-10 (Estimated); Study Completion 2021-10 (Estimated)

PRIMARY OUTCOMES:
Recurrence of Atrial Fibrillation | 12 Months
  Recurrence of atrial fibrillation will be defined by detection of an episode of atrial fibrillation, atrial flutter or atrial tachycardia lasting for more than 30 seconds during any of the study follow-up periods up to one year post-ablation.

SECONDARY OUTCOMES:
Recurrence of Atrial Fibrillation Stratified by Atrial Fibrillation Type | 12 Months
  Recurrence of atrial fibrillation type will be compared to historical data of ablations targeting only pulmonary vein isolation

CONTACTS AND LOCATIONS:
Overall Officials: Nassir F Marrouche, M.D., Principal Investigator — University of Utah

IPD SHARING:
Plan to Share IPD: No